CLINICAL TRIAL: NCT04260711
Title: The Safety and Cost-effectiveness of Discontinuing Disease-modifying Therapies in Stable Relapsing - Onset Multiple Sclerosis (DOT-MS): a Randomized Rater-blinded Multicenter Trial.
Brief Title: Discontinuing Disease-modifying Therapies in Stable Relapsing - Onset Multiple Sclerosis (DOT-MS).
Acronym: DOT-MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Eline Coerver, Corresponding investigator, (also: E.M.M. Strijbis (coordinating investigator) and J. Killestein (principal investigator)), Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL71260.029.19
Record Dates: First submitted 2020-01-21; First posted 2020-02-07 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: multiple sclerosis; disease modifying therapy
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Interferons; Glatiramer Acetate; Dimethyl Fumarate; teriflunomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation of DMT (Experimental): Discontinuation of first-line disease modifying therapy (any of the interferons, glatiramer acetate, dimethylfumarate, teriflunomide)
  Interventions: Drug: DMT
- Continuation of DMT (No Intervention): Continuation of first-line disease modifying therapy (any of the interferons, glatiramer acetate, dimethylfumarate, teriflunomide)

INTERVENTIONS:
Drug: DMT — Discontinuation of patients' own disease modifying therapy (any of the interferons, glatiramer acetate, dimethylfumarate, teriflunomide)
  Other Names: Interferon; Glatiramer acetate; Dimethylfumarate; Teriflunomide
  Arms: Discontinuation of DMT

SUMMARY:
The aim of this study is to identify whether it is possible to safely discontinue treatment in relapsing-onset MS patients who have shown no evidence of active inflammation in the years prior to inclusion clinically and/or radiologically. The secondary objectives address the questions whether the discontinuation of first-line treatment has an effect on disability progression and whether the discontinuation of first-line treatment improves the quality of life for the patient. Furthermore, blood collections will be included to assess whether it is possible to retrospectively predict possible return of inflammatory activity with biomarkers such as neurofilament light (NFL) or patient characteristics such as disease activity prior to disease modifying therapy (DMT). In case of emerging disease activity after the cessation of therapy we will assess if reinitiation will lead to NEDA again, and if there are long-term consequences. If possible, post-hoc analysis are performed for the different types of treatment compounds.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local privacy regulations.
* Definite diagnosis of relapsing-onset MS according to the revised McDonald 2017 criteria
* Treatment with one of the first-line DMTs: any of the interferons, glatiramer acetate, dimethylfumarate, teriflunomide
* Complete absence of inflammatory activity (no objectively defined and confirmed relapses, no significant number (2 or more) of new-T2 lesions and no contrast-enhancing lesions) for 5 consecutive years under first-line treatment

Exclusion Criteria:

* A switch between first-line disease modifying therapy over two years prior to inclusion, in case the switch has been due to in effectivity of the first DMT.
* Women who want to discontinue medication because of a pregnancy wish and women who are pregnant or expect to become pregnant during the study period
* Patients that have previously used interferon-beta and have been tested positive for neutralizing antibodies (NAbs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical relapses | 2 years
  New clinically confirmed relapses (defined according to the definition most often used in MS phase-III trials: the onset of new or recurrent symptoms that last > 24 hours, that are accompanied by new objective abnormalities on a neurological examination and that are not explained by non-MS processes such as fever, infection, severe stress or drug toxicity).
New lesions on MRI-brain | 2 years
  New inflammatory disease activity on MRI (defined as 3 or more lesions on T2-weighted vimages or 2 or more gadolinium enhancing lesions on T1-weighted post-contrast MRI).

SECONDARY OUTCOMES:
EDSS (Expanded Disability Status Scale) | 2 years
  This score indicates disability on a scale of 0 to 10. A higher score indicates more disability.
9-hole peg test | 2 years
  9-hole peg test (9HPT): test on hand function, measured in seconds. A shorter time indicates a better hand function.
Timed 25-Foot Walk | 2 years
  Timed 25-foot walk (T25FW): walking test, measured in seconds. A shorter time indicates a better walking function.
Symbol Digits Modalities Test | 2 years
  Symbol Digits Modalities Test (SDMT): measures cognition. Scored with a number from 0 to 110, a higher score indicates better cognitive function.
MRI-parameter: T1 post-contrast lesion number | 2 years
  Number of lesions on T1 post-contrast MRI
MRI-parameter: T2 post-contrast lesion number | 2 years
  Number of lesions on T2-MRI
Multiple Sclerosis Impact Scale (MSIS-29) | 2 years
  Questionnaire on the impact of MS on day-to-day life
Short Form health survey (SF-36) | 2 years
  Questionnaire on general health
Checklist Individual Strength (CIS20r) | 2 years
  Questionnaire on fatigue
Treatment Satisfaction Questionnaire for Medication (TSQM) | 2 years
  Questionnaire on treatment satisfaction
EuroQol 5 dimensions questionnaire (EQ-5D-5L) | 2 years
  Questionnaire on quality of life and costs
Medical consumption questionnaire (iMCQ) | 2 years
  Questionnaire on medical consumption
Productivity costs questionnaire (iPCQ) | 2 years
  Questionnaire on productivity
Neurofilament light level in serum | 2 years
  Neurofilament light levels in serum

CONTACTS AND LOCATIONS:
Overall Officials: J. Killestein, prof. dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coerver EME, Fung WH, de Beukelaar J, Bouvy WH, Canta LR, Gerlach OHH, Hoitsma E, Hoogervorst ELJ, de Jong BA, Kalkers NF, van Kempen ZLE, Lovenich H, van Munster CEP, van Oosten BW, Smolders J, Vennegoor A, Zeinstra EMPE, Barrantes-Cepas M, Kooij G, Schoonheim MM, Lissenberg-Witte BI, Teunissen CE, Moraal B, Barkhof F, Uitdehaag BMJ, Mostert J, Killestein J, Strijbis EMM. Discontinuation of First-Line Disease-Modifying Therapy in Patients With Stable Multiple Sclerosis: The DOT-MS Randomized Clinical Trial. JAMA Neurol. 2025 Feb 1;82(2):123-131. doi: 10.1001/jamaneurol.2024.4164. PMID 39652340